CLINICAL TRIAL: NCT02167308
Title: Effect of Laser Acupuncture on Obesity: a Patient-Assessor-Blinded, Randomized, Sham-controlled Crossover Trial
Brief Title: Effect of Laser Acupuncture on Obesity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Chi-chuan Tseng, MD, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 103-1403A3
Record Dates: First submitted 2014-06-14; First posted 2014-06-19 (Estimated); Last update posted 2014-06-19 (Estimated); Status verified 2014-06

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Laser acupuncture group (Active Comparator): Subjects will receive 24 activated laser acupuncture treatments. The laser will be applied for 10 seconds to each of the selected acupuncture points.
  Interventions: Device: Laser acupuncture
- Control group (Sham Comparator): Subjects in the control group will undergo sham laser acupuncture treatment with no laser power output. Acupuncture points, application duration, and total number of treatments will be identical to the Laser acupuncture group.
  Interventions: Device: Laser acupuncture

INTERVENTIONS:
Device: Laser acupuncture — a GaAlAs semiconductor diode Laser Phototherapy Device with a wavelength of 808nm. Maximum power output is 150 milliwatt in continuous wave mode.

SUMMARY:
Background: Obesity-related diseases have a profound economic impact on health care systems. Laser acupuncture has been shown to have beneficial effects on obesity. However, to our knowledge, those trials were either non-randomized, non-blinded, or included low-calorie diet control. Investigators have therefore designed a patient-assessor-blinded, randomized, sham-controlled crossover trial to investigate the significance of laser acupuncture on obesity.

Methods/design: One hundred and four subjects above 20 years of age with a body mass index (BMI) of over 25 kg/m2 will be divided into two groups: experimental and control. Each subject will receive the treatment relevant to their group three times a week for eight weeks. After eight weeks of treatment the subject will enter a two week washout period, after which the subjects will switch groups. Measurements will include BMI, body fat percentage, waist-to-hip ratio (WHR), waist circumference, hip circumference, skinfold thickness, thigh circumference, body fat, blood pressure, heart rate, hunger, and the 36-item short-form health survey (SF-36).

Discussion: The results of this pilot study will provide the basis for future large-scale multicenter trials investigating the effects of laser acupuncture on obesity.

DETAILED DESCRIPTION:
The number of obese people around the world has been increasing rapidly. It has been estimated that over 10% of the world's adult population are obese. Obesity is associated with increased risk of coronary heart disease, type II diabetes, stroke, osteoarthritis, and certain types of cancer. These deleterious conditions are detrimental to individuals' quality of life, and places emotional and financial burden on the individual, their families, and society as a whole. Much more needs to be done to improve treatments for obesity.

Current methods to treat obesity include dietary intervention, lifestyle intervention, drug intervention, or bariatric surgery. Among these, acupuncture, in a comprehensive program for weight loss, has been increasing in popularity. However, previous systematic reviews assessing the effects of acupuncture on obesity discovered promising but inconclusive results. The low quality methodology used in those trials further reduced the strength of those conclusions. In addition, the lack of safety procedures used in traditional manual acupuncture could lead to adverse events such as retroperitoneal abscess, rapid dermal spread of breast cancer, pneumothorax, cardiac tamponade, viral hepatitis, and granuloma.

In comparison with traditional manual acupuncture, laser acupuncture therapy has several advantages. These advantages include ease of application, precision in dose measurement, painlessness, and non-invasiveness. It is a quick and safe therapy with low cost and no risk of infection. As laser acupuncture does not produce local sensation, double blind randomized controlled studies are also much easier to perform.

Laser acupuncture has been widely used in medical fields for over 30 years. Clinical research on the efficacy of laser acupuncture has also increased. Several studies have showed that laser acupuncture could be an effective treatment of obesity. Low-level laser therapy as a non-invasive approach for body contouring and spot fat reduction has also been reported. However, there are several experimental limitations that have to be considered. For instance, absence of placebo (sham) control, combination with low-calorie diet, and lack of sufficient comparative parameters have been questioned . For these reasons, investigators decided to conduct a patient-assessor-blinded, randomized, sham-controlled crossover pilot trial to investigate the effects of laser acupuncture with Gallium Aluminum Arsenide (GaAlAs) laser irradiation on weight loss, fat reduction, body contouring, and quality of life in people suffering from obesity.

ELIGIBILITY:
Inclusion Criteria:

* Individuals are eligible if they are above 20 years of age and have a BMI over 25 kg/m2. BMI cutoffs were adopted from a proposed classification of weight by BMI in adult Asians, including the obese I (BMI: 25-29.9 kg/m2) and obese II (BMI ≥30 kg/m2) categories.

Exclusion Criteria:

* cardiovascular disease
* diabetes
* endocrine abnormalities
* renal disease
* contagious skin condition
* epilepsy
* tumor
* mental disorder
* pregnant
* photosensitivity reactions to laser treatment
* uses a pacemaker
* used medications known to affect one's weight up to one month in advance
* un-willing to comply with the study protocol

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2014-06; Primary Completion 2016-07 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
BMI change from baseline | week 26

SECONDARY OUTCOMES:
Body fat percentage | week 26
Waist-to-Hip ratio (WHR) | week 26
Hunger | week 26
  For hunger, a Visual Analogue Scale (VAS) with horizontal lines will be used, graded from 0 mm, representing no hunger, to 100 mm, representing the most extreme hunger imaginable. Subjects will be asked to mark their level of hunger on the VAS.
Quality of life | week 26
  Will be assessed via validated questionnaire (short-form 36-item Health Survey, SF36)

OTHER OUTCOMES:
Skin fold thickness | week 26
Thigh circumference | week 26
Blood pressure | week 26
Heart rate | week 26

CONTACTS AND LOCATIONS:
Overall Officials: Chi-Chuan Tseng, MD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Chiayi County, Taiwan

REFERENCES:
- [Derived] Tseng CC, Tseng A, Chang CH. Effect of laser acupuncture on obesity: study protocol for a randomized controlled trial. Trials. 2015 May 15;16:217. doi: 10.1186/s13063-015-0748-4. PMID 25972018